CLINICAL TRIAL: NCT01801631
Title: Tailored Support for Type 2 Diabetes Patients With an Acute Coronary Event After Discharge From Hospital
Acronym: Diacourse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Prof. G.E.H.M. Rutten, Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DF2009-70; Dutch trial registration (Registry Identifier: NTR3076)
Record Dates: First submitted 2013-02-14; First posted 2013-03-01 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes; Acute Coronary Event
Keywords: Type 2 diabetes; Acute Coronary Event (ACE); Distress; Self-efficacy; Quality of Life; Depression; Primary care; Illness representations
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression | interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home visits (Experimental): In addition to usual care the patients will receive three home visits from a trained diabetes nurse. The first visit (65 minutes) is within three weeks after discharge from the hospital; the second visit (45 minutes) is two weeks later and the third visit (45 minutes) is two months after the second home visit.
  Interventions: Other: Home visits
- Consultation by telephone (Other): In addition to usual care patients will receive a consultation by telephone within three weeks after discharge to offer them personal attention. In this consultation they will get the opportunity to discuss in ten to fifteen minutes how they feel in the period after discharge.
  Interventions: Other: Consultation by telephone

INTERVENTIONS:
Other: Home visits — In addition to usual care the patients will receive three home visits from a trained diabetes nurse. The first visit (65 minutes) is within three weeks after discharge from the hospital; the second visit (45 minutes) is two weeks later and the third visit (45 minutes) is two months after the second home visit.
  Arms: Home visits
Other: Consultation by telephone — In addition to usual care patients will receive a consultation by telephone within three weeks after discharge to offer them personal attention. In this consultation they will get the opportunity to discuss in ten to fifteen minutes how they feel in the period after discharge.
  Arms: Consultation by telephone

SUMMARY:
Background: In type 2 diabetes mellitus patients, an acute coronary event (ACE) may result in a decreased quality of life and increased distress. According to the American Diabetes Association, transition from the acute care setting is a high-risk time for all patients, but tailored support specific to diabetes is scarce in that period. The investigators developed an intervention by a diabetes nurse to help diabetic patients reduce distress after their first ACE. The intervention is based on Bandura's Social Cognitive Theory, Leventhal's Common Sense Model, and on results of focus groups which were conducted to define the needs and wishes of type 2 diabetes patients and their partners regarding professional support after an ACE. The aim of this study is to evaluate the effectiveness of the intervention to reduce distress. The hypothesis is that patients who receive the intervention will have less diabetes related distress compared to the control group.

Methods/Design: Randomized controlled trial. Patients will be recruited directly after discharge from hospital. A diabetes nurse will visit the patients in the intervention group (n = 100) within three weeks after discharge from hospital, two weeks later and two months later. The control group (n = 100) will receive a telephone consultation. The primary outcome is diabetes related distress, measured with the Problem Areas in Diabetes questionnaire (PAID). Secondary outcomes are quality of life, anxiety, depression, HbA1c, blood pressure and lipids. Mediating variables are self-management, self-efficacy and illness representations. Variables will be measured with questionnaires directly after discharge from hospital and five months later. Biomedical variables will be obtained from the records from the primary care physician and the hospital. Differences between groups in change over time will be analyzed according to the intention-to-treat principle.

Discussion: Type 2 diabetes patients who experience a first ACE need tailored support after discharge from the hospital. This trial will provide evidence of the effectiveness of a supportive intervention to reduce distress in these patients.

DETAILED DESCRIPTION:
See citation design paper

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes (>1 year)
* Discharged from the hospital after a first acute coronary event defined as a Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG) procedure or Percutaneous Transluminal Coronary Angioplasty (PTCA)
* Sufficient knowledge of the Dutch language

Exclusion Criteria:

* A serious illness or condition which will prevent full participation
* Not able to fill in questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes related distress | At 2 weeks and 5 months after discharge from hospital
  Diabetes related distress measure with the Problem Areas in Diabetes (PAID) questionnaire. The PAID is a Self-reported questionnaire consisting of twenty statements identified as common negative emotions related to living with diabetes. Each item is rated on a 5-point Likert scale, ranging from 0 ("not a problem") to 4 ("a serious problem"). The total score is transformed to a 0-100 scale, with higher score representing higher distress.

SECONDARY OUTCOMES:
Change in Well-being | At 2 weeks and 5 months after discharge from hospital
  Measured with the WHO-Five Well-being Index (WHO-5). The five items covering positive mood (good spirits, relaxation), vitality (being active and waking up fresh and rested), and general interests (being interested in things) in the past two weeks
Change in Quality of life | At 2 weeks and 5 months after discharge from hospital
  Euroqol 5 Dimensions (EQ-5D) and the Euroqol Visual Scale (EQ-VAS). The EQ-5D measures general health status on five dimensions:
  1. Mobility
  2. Self-care
  3. Usual activities
  4. Pain/discomfort
  5. Anxiety/depression The EQ-VAS measures the overall health state on a graded, vertical line.
Change in Anxiety and depression | At 2 weeks and 5 months after discharge from hospital
  Measured with the Hospital Anxiety and Depression Scale (HADS). A questionnaire measuring anxiety (7 items) and depression (7 items).
Change in Physical activity | At 2 weeks and 5 months after discharge from hospital
  Measured with the International Physical Activity Questionnaire (IPAQ). 29 Items measure how many days' physical activities are performed during the past seven days in four domains (work, transportation, housework and leisure-time).
Change in Self care | At 2 weeks and 5 months after discharge from hospital
  Measured with the Summary of the Diabetes Self-Care Activities Measure (SDSCA). Eleven items assessing several aspects of the diabetes regimen: general diet, specific diet, exercise, blood glucose testing, foot care, and smoking. Items measure how many days a patient has performed self-care activities in the last seven days.
Change in Diabetes coping | At 2 weeks and 5 months after discharge from hospital
  Measured with the Diabetes Coping Measure (DCM) consisting of four scales measuring diabetes coping: tackling spirit, avoidance, passive resignation and diabetes integration.
Change in Biomedical variables | At 2 weeks and 5 months after discharge from hospital
  Blood pressure, blood lipids (total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides) and body mass index

OTHER OUTCOMES:
Change in Self-efficacy | At 2 weeks and 5 months after discharge from hospital
  Measured with the Confidence in Diabetes Self-care questionnaire consisting of 20 items measuring diabetes specific self-efficacy.
Change in Illness perceptions | At 2 weeks and 5 months after discharge from hospital
  Measured with the Illness Perception Questionnaire (IPQ) - short version. Questionnaire assessing the cognitive representation of illness, focuses on seven scales, assessing (1) Timeline acute/chronic and (2) Timeline cyclical (3) Consequences (4) Personal control (5) Treatment control (6) Illness coherence (7) Emotional representation
Change in Spousal support | At 2 weeks and 5 months after discharge from hospital
  Measured with the Active Engagement, Protective Buffering and Overprotection (ABO) questionnaire. Five items measure active engagement, eight items measure protective buffering and six items measure overprotection

CONTACTS AND LOCATIONS:
Overall Officials: Guy E. Rutten, Professor, Principal Investigator — UMC Utrecht
Locations (13):
- Netherlands (13):
  - Meander Medical Center, Amersfoort
  - Gelre Hospitals, Apeldoorn
  - Lievensberg Hospital, Bergen op Zoom
  - Amphia Hospital, Breda
  - Gemini Hospital, Den Helder
  - Admiraal de Ruyter Hospital, Goes
  - Beatrix Hospital, Gorinchem
  - Westfriesgasthuis, Hoorn
  - Sint Antonius Hospital, Nieuwegein
  - Canisius Wilhelmina Hospital, Nijmegen
  - Diakonessenhuis, Utrecht
  - Sint Antonius Hospital, Utrecht
  - University Medical Center, Utrecht

REFERENCES:
- [Background] Kasteleyn MJ, Gorter KJ, Stellato RK, Rijken M, Nijpels G, Rutten GE. Tailored support for type 2 diabetes patients with an acute coronary event after discharge from hospital - design and development of a randomised controlled trial. Diabetol Metab Syndr. 2014 Jan 18;6(1):5. doi: 10.1186/1758-5996-6-5. PMID 24438342
- [Background] Kasteleyn MJ, Gorter KJ, van Puffelen AL, Heijmans M, Vos RC, Jansen H, Rutten GE. What follow-up care and self-management support do patients with type 2 diabetes want after their first acute coronary event? A qualitative study. Prim Care Diabetes. 2014 Oct;8(3):195-206. doi: 10.1016/j.pcd.2013.12.001. Epub 2014 Jan 3. PMID 24389352